CLINICAL TRIAL: NCT02234752
Title: A Proof-of Concept Trial of Galantamine and Memantine for Cognitive Impairments in Schizophrenia: Is the Combination Effective?
Brief Title: Galantamine and Memantine Combination for Cognitive Impairments in Schizophrenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding no longer available and PI no longer working at the institution
Sponsor: Sheppard Pratt Health System (Other)
Responsible Party: Principal Investigator, Maju Koola, Principal Investigator, Sheppard Pratt Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHS IRB # 604148-4
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2016-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Cognition; Cognitive Impairment; Galantamine; Memantine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognitive Dysfunction | interventions — Galantamine; Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Galantamine ER, Memantine XR (Experimental): Week 1, Galantamine ER 8 mg HS & Memantine XR 7 mg HS Week 2, Galantamine ER 16 mg HS & Memantine XR 14 mg HS Weeks 3-6, Galantamine ER 24 mg HS & Memantine XR 21 mg HS
  Interventions: Drug: Galantamine ER; Drug: Memantine XR

INTERVENTIONS:
Drug: Galantamine ER
  Other Names: Razadyne; Razadyne ER; Formerly known as Reminyl
Drug: Memantine XR
  Other Names: Namenda

SUMMARY:
Aim: To examine the efficacy of the combination of galantamine and memantine for the treatment of cognitive deficits in outpatients with schizophrenia.

Hypothesis: A combination of galantamine and memantine will improve cognitive impairments in patients with schizophrenia.

This is an open-label study to evaluate whether a six week course of galantamine ER and memantine XR is effective in improving the cognitive performance of patients with schizophrenia or schizoaffective disorder. The primary outcome measure will be the change in level of cognition as measured by the MATRICS Consensus Cognitive Battery (MCCB). The results of the MATRICS collaborative project recommended the need for standardized cognitive tests that better distinguish the different facets of cognitive dysfunction in schizophrenia. The MCCB will assess the following seven domains: attention/vigilance, reasoning and problem solving, processing speed, social cognition, verbal learning and memory, visual learning and memory, and working memory. The MCCB will be administered at baseline and at the end of the study. We will report total score and each domain score in the MCCB at baseline and six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female aged 18 to 55 years (inclusive).
* Have a DSM-5 diagnosis of schizophrenia or schizoaffective disorder confirmed by medical records. Duration of illness must be ≥ 1year.
* Be clinically stable for at least two months (i.e., has no more than a "moderately severe" severity rating on the following BPRS items: hallucination, unusual thought content and conceptual disorganization.
* Have not had a psychiatric hospitalization in the two months prior to screening.
* Be taking any 1st generation antipsychotic prescribed in the absence of a concomitant anticholinergic or 2nd generation antipsychotic and minimal extrapyramidal symptoms
* Have a Simpson-Angus Score (SAS) < 6
* Be on current medication regimen for at least six weeks before screening at stable dose and frequency for at least 30 days before screening.
* Be in good general health and expected to complete the clinical study as designed.
* Subjects of childbearing potential must agree to use two forms of non-hormonal contraception (dual contraception) consistently during the screening and treatment periods of the trial, and for 30 days after the final dose of the study medications.
* Females of child-bearing potential must have a negative urine pregnancy test at baseline. This may also be done at subsequent visits if subject reports possibility of pregnancy.
* Have a negative urine drug screen at screening. This may be repeated at the discretion of the primary investigator.
* Have adequate hearing, vision, and language skills to perform the procedures specified in the protocol.
* Be capable of providing informed consent and have voluntarily provided informed consent.

Exclusion Criteria:

* Have an active, clinically significant unstable medical condition with 30 days prior to screening.
* Have dementia.
* Are pregnant, breastfeeding, or planning to become pregnant
* Are taking or thinking about taking oral contraceptives or an injectable contraceptive.
* Are taking benztropine at a dose greater than 2 mg daily.
* Have a history of Pervasive Development Disorder.
* Have a history of significant head injury/trauma (defined by one of more of the following: loss of consciousness for more than one hour; recurring seizures resulting from the head injury; and/or clear cognitive sequelae of the injury requiring cognitive rehabilitation.)
* Have an allergy to anticholinesterase medications (galantamine, rivastigimine, donepezil) and memantine
* Have a DSM-5 diagnosis of alcohol and/or substance use disorder (other than caffeine and tobacco) within the last 6 months.
* Are taking a restricted medication: Amitriptyline, Doxepin, Imipramine, Flexeril, Clozapine, and/or cortisol (any oral, injectable, or topical steroid medication)
* Have a history of seizures excluding a childhood febrile seizure
* Have received ECT within the last three months prior to screening.
* Have participated in a clinical trial of any other psychotropic medication within last two months prior to screening.
* Have a "severe" or "extremely severe" severity rating on the BPRS items: hallucination or unusual thought content.
* Have more than a "moderate" severity rating on the BPRS item conceptual disorganization .
* Are currently taking 3 or more antipsychotic medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maju M. Koola, MD, Principal Investigator — Sheppard Pratt Health System
Locations (1):
- Sheppard Pratt Health System, Baltimore, Maryland, United States

REFERENCES:
- [Background] Koola MM, Buchanan RW, Pillai A, Aitchison KJ, Weinberger DR, Aaronson ST, Dickerson FB. Potential role of the combination of galantamine and memantine to improve cognition in schizophrenia. Schizophr Res. 2014 Aug;157(1-3):84-9. doi: 10.1016/j.schres.2014.04.037. Epub 2014 May 28. PMID 24878431
- [Background] Koola MM. Kynurenine pathway and cognitive impairments in schizophrenia: Pharmacogenetics of galantamine and memantine. Schizophr Res Cogn. 2016 Jun;4:4-9. doi: 10.1016/j.scog.2016.02.001. PMID 27069875
- [Result] Koola MM, Sklar J, Davis W, Nikiforuk A, Meissen JK, Sawant-Basak A, Aaronson ST, Kozak R. Kynurenine pathway in schizophrenia: Galantamine-memantine combination for cognitive impairments. Schizophr Res. 2018 Mar;193:459-460. doi: 10.1016/j.schres.2017.07.005. Epub 2017 Jul 11. No abstract available. PMID 28705532

RESULTS

PARTICIPANT FLOW:
Groups:
- Galantamine ER, Memantine XR: Week 1, Galantamine ER 8 mg HS & Memantine XR 7 mg HS Week 2, Galantamine ER 16 mg HS & Memantine XR 14 mg HS Weeks 3-6, Galantamine ER 24 mg HS & Memantine XR 21 mg HS
  Galantamine ER
  Memantine XR
Period: Overall Study
Arm/Group | Galantamine ER, Memantine XR
Started | 3
Completed | 2
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Galantamine ER, Memantine XR
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Level of Cognition
Description: The primary outcome measure will be the change in level of cognition as measured by the MATRICS Consensus Cognitive Battery (MCCB). In schizophrenia, usual composite scores are 20-39. In healthy controls, usual composite scores are normalized to 40-60. Higher values of composite scores mean better cognition. Test scores are normalized to healthy controls, therefore no min-max range is available. Final scores calculated by MATRICS Consensus Cognitive Battery software. Exact minimum/maximum are not known to provider. Overall composite scores are reported.
Time Frame: Baseline and 6-Weeks
Population: Participant 3 only provided baseline data
Measure: Number; unit: units on a scale
Arm/Group | Galantamine ER, Memantine XR
Number analyzed (Participants) | 3
units on a scale
  Baseline Participant 1: number analyzed (Participants) | 1
  Baseline Participant 1 | 48
  Week 6 Participant 1: number analyzed (Participants) | 1
  Week 6 Participant 1 | 48
  Baseline Participant 2: number analyzed (Participants) | 1
  Baseline Participant 2 | 32
  Week 6 Participant 2: number analyzed (Participants) | 1
  Week 6 Participant 2 | 25
  Baseline Participant 3: number analyzed (Participants) | 1
  Baseline Participant 3 | 9

2. Secondary Outcome: Free Tryptophan (TRP)
Description: The secondary outcome measure will be change in metabolite values. Values were collected in triplicate.
Time Frame: Baseline and 6-Weeks
Population: Participant 3 only provided baseline data
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | KP Metabolites Values
Number analyzed (Participants) | 3
µM
  Baseline tryptophan Participant 1: number analyzed (Participants) | 1
  Baseline tryptophan Participant 1 | 51.94 (2.39)
  Week-6 tryptophan Participant 1: number analyzed (Participants) | 1
  Week-6 tryptophan Participant 1 | 55.72 (2.83)
  Baseline tryptophan Participant 2: number analyzed (Participants) | 1
  Baseline tryptophan Participant 2 | 32.17 (1.05)
  Week-6 tryptophan Participant 2: number analyzed (Participants) | 1
  Week-6 tryptophan Participant 2 | 24.96 (1.33)
  Baseline tryptophan Participant 3: number analyzed (Participants) | 1
  Baseline tryptophan Participant 3 | 35.07 (1.22)

3. Secondary Outcome: Kynurenic Acid (KYNA)
Description: The secondary outcome measure will be change in metabolite values. Values were collected in triplicate. MS* AUC is mass spectrometry times area under the curve.
Time Frame: Baseline and 6-Weeks
Population: Participant 3 only provided baseline data
Measure: Mean (Standard Deviation); unit: MS* AUC
Arm/Group | KP Metabolites Values
Number analyzed (Participants) | 3
MS* AUC
  Baseline KYNA Participant 1: number analyzed (Participants) | 1
  Baseline KYNA Participant 1 | 103911 (20870)
  Week-6 KYNA Participant 1: number analyzed (Participants) | 1
  Week-6 KYNA Participant 1 | 83737 (25309)
  Baseline KYNA Participant 2: number analyzed (Participants) | 1
  Baseline KYNA Participant 2 | 95139 (36663)
  Week-6 KYNA Participant 2: number analyzed (Participants) | 1
  Week-6 KYNA Participant 2 | 73280 (15567)
  Baseline KYNA Participant 3: number analyzed (Participants) | 1
  Baseline KYNA Participant 3 | 93163 (41519)

4. Secondary Outcome: Kynurenine (KYN)
Description: The secondary outcome measure will be change in metabolite values. Values were collected in triplicate.
Time Frame: Baseline and 6-Weeks
Population: Participant 3 only provided baseline data
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | KP Metabolites Values
Number analyzed (Participants) | 3
µM
  Baseline KYN Participant 1: number analyzed (Participants) | 1
  Baseline KYN Participant 1 | 1.62 (0.12)
  Week-6 KYN Participant 1: number analyzed (Participants) | 1
  Week-6 KYN Participant 1 | 1.85 (0.24)
  Baseline KYN Participant 2: number analyzed (Participants) | 1
  Baseline KYN Participant 2 | 0.86 (0.13)
  Week-6 KYN Participant 2: number analyzed (Participants) | 1
  Week-6 KYN Participant 2 | 0.71 (0.05)
  Baseline KYN Participant 3: number analyzed (Participants) | 1
  Baseline KYN Participant 3 | 0.76 (0.04)

5. Secondary Outcome: Picolinic Acid (PIC)
Description: as for outcome 3
Time Frame: Baseline and 6-Weeks
Population: Participant 3 only provided baseline data
Measure: Mean (Standard Deviation); unit: MS* AUC
Arm/Group | KP Metabolites Values
Number analyzed (Participants) | 3
MS* AUC
  Baseline PIC Participant 1: number analyzed (Participants) | 1
  Baseline PIC Participant 1 | 44021 (4470)
  Week-6 PIC Participant 1: number analyzed (Participants) | 1
  Week-6 PIC Participant 1 | 29542 (383)
  Baseline PIC Participant 2: number analyzed (Participants) | 1
  Baseline PIC Participant 2 | 81883 (7344)
  Week-6 PIC Participant 2: number analyzed (Participants) | 1
  Week-6 PIC Participant 2 | 63745 (1535)
  Baseline PIC Participant 3: number analyzed (Participants) | 1
  Baseline PIC Participant 3 | 40189 (4342)

6. Secondary Outcome: KYN/TRP
Description: The secondary outcome measure will be change in metabolite values. Values were collected in triplicate. AUC ratio reported.
Time Frame: Baseline and 6-Weeks
Population: Participant 3 only provided baseline data
Measure: Number; unit: AUC Ratio
Arm/Group | KP Metabolites Values
Number analyzed (Participants) | 3
AUC Ratio
  Baseline KYN/TRP Participant 1: number analyzed (Participants) | 1
  Baseline KYN/TRP Participant 1 | 1.21
  Week-6 KYN/TRP Participant 1: number analyzed (Participants) | 1
  Week-6 KYN/TRP Participant 1 | 1.31
  Baseline KYN/TRP Participant 2: number analyzed (Participants) | 1
  Baseline KYN/TRP Participant 2 | 1.06
  Week-6 KYN/TRP Participant 2: number analyzed (Participants) | 1
  Week-6 KYN/TRP Participant 2 | 0.8
  Baseline KYN/TRP Participant 3: number analyzed (Participants) | 1
  Baseline KYN/TRP Participant 3 | 0.79

7. Secondary Outcome: KYNA/KYN
Description: as for outcome 6
Time Frame: Baseline and 6-Weeks
Population: Participant 3 only provided baseline data
Measure: Number; unit: AUC Ratio
Arm/Group | KP Metabolites Values
Number analyzed (Participants) | 3
AUC Ratio
  Baseline KYNA/KYN Participant 1: number analyzed (Participants) | 1
  Baseline KYNA/KYN Participant 1 | 0.075
  Week-6 KYNA/KYN Participant 1: number analyzed (Participants) | 1
  Week-6 KYNA/KYN Participant 1 | 0.050
  Baseline KYNA/KYN Participant 2: number analyzed (Participants) | 1
  Baseline KYNA/KYN Participant 2 | 0.121
  Week-6 KYNA/KYN Participant 2: number analyzed (Participants) | 1
  Week-6 KYNA/KYN Participant 2 | 0.114
  Baseline KYNA/KYN Participant 3: number analyzed (Participants) | 1
  Baseline KYNA/KYN Participant 3 | 0.152

8. Secondary Outcome: PIC/KYN
Description: as for outcome 6
Time Frame: Baseline and 6-Weeks
Population: Participant 3 only provided baseline data
Measure: Number; unit: AUC Ratio
Arm/Group | KP Metabolites Values
Number analyzed (Participants) | 3
AUC Ratio
  Baseline PIC/KYN Participant 1: number analyzed (Participants) | 1
  Baseline PIC/KYN Participant 1 | 0.0317
  Week-6 PIC/KYN Participant 1: number analyzed (Participants) | 1
  Week-6 PIC/KYN Participant 1 | 0.0175
  Baseline PIC/KYN Participant 2: number analyzed (Participants) | 1
  Baseline PIC/KYN Participant 2 | 0.1039
  Week-6 PIC/KYN Participant 2: number analyzed (Participants) | 1
  Week-6 PIC/KYN Participant 2 | 0.0989
  Baseline PIC/KYN Participant 3: number analyzed (Participants) | 1
  Baseline PIC/KYN Participant 3 | 0.0655

ADVERSE EVENTS:
Arm/Group | Galantamine ER, Memantine XR
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galantamine ER, Memantine XR (N=3)
Increased tiredness (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Lightheadedness (General disorders) | 1 (3)
Dizziness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No